CLINICAL TRIAL: NCT05219968
Title: ENLIGHTEN 1: A Phase III, Randomized, Blinded, Controlled, Parallel-Group Trial to Evaluate the Efficacy and Safety of LYR-210 for the Treatment of Chronic Rhinosinusitis (CRS) in Adults
Brief Title: Efficacy and Safety of LYR-210 for the Treatment of Chronic Rhinosinusitis in Adults
Acronym: ENLIGHTEN 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lyra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYR-210-2021-004
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Sinusitis; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYR-210 (Experimental): Single administration of LYR-210 drug matrix (7500 μg)
  Interventions: Drug: LYR-210; Other: Background Therapy
- Sham procedure control (Sham Comparator): Single mock administration procedure
  Interventions: Drug: Sham procedure control; Other: Background Therapy

INTERVENTIONS:
Drug: LYR-210 — LYR-210 drug matrix (mometasone furoate)
  Arms: LYR-210
Drug: Sham procedure control — Sham procedure control
  Arms: Sham procedure control
Other: Background Therapy — Daily Saline Irrigation

SUMMARY:
Multicenter, phase III, randomized, blinded, controlled, parallel group with safety extension phase with crossover or continued treatment.

DETAILED DESCRIPTION:
This is a 52-week, multicenter, phase III, randomized, blinded, controlled, parallel group with a 24-week treatment period followed by a safety extension phase with crossover or continued treatment to evaluate the efficacy and safety of LYR-210 compared with sham control for treatment in adults with CRS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Diagnosed as having CRS
* Undergone at least 2 trials of medical treatments in the past
* Mean 3 cardinal symptom (3CS) score
* Bilateral ethmoid disease confirmed on CT
* Has been informed of the nature of the study and provided written informed consent
* Agrees to comply with all study requirements
* If on a waiting list for sinonasal surgery, willing to be removed from list or have surgery date cancelled for the duration of the study.

Exclusion Criteria:

* Inability to tolerate topical anesthesia or endoscopic procedure
* Previous nasal surgery
* Presence of nasal polyp grade 2 or higher
* Seasonal allergic rhinitis
* Perennial rhinitis with symptoms that are well controlled by regular use of intranasal corticosteroids
* Severe asthma
* History or clinical evidence or suspicion of invasive fungal sinusitis, allergic fungal rhinosinusitis, atrophic rhinitis, or odontogenic sinusitis
* Obstruction preventing proper placement and retention of LYR-210 as seen on endoscopy
* Anatomic variation that, in the opinion of the investigator, would adversely impact placement of LYR-210 as seen on CT
* Known history of hypersensitivity or intolerance to corticosteroids
* Known history of hypothalamic pituitary adrenal axial dysfunction
* Previous pituitary or adrenal surgery
* Dental procedure/implant on maxillary dentition within 4 weeks of the Screening visit.
* Past or present acute or chronic intracranial or orbital complications of CRS
* History or diagnosis (in either eye) of glaucoma or ocular hypertension
* Past or present functional vision in only 1 eye
* Past, present, or planned organ transplant or chemotherapy with immunosuppression
* Currently positive for COVID-19 or residual sinonasal symptoms from a previous COVID-19 infection
* Pregnant or breast feeding. Females of child-bearing potential must test negative for pregnancy at the time of screening
* Evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments
* Currently participating in an investigational drug or device study
* Determined by the investigator as not suitable to be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (24):
  - Lyra Investigational Site, Birmingham, Alabama
  - Lyra Investigational Site, Escondido, California
  - Lyra Investigational Site, La Mesa, California
  - Lyra Investigational Site, Sacramento, California
  - Lyra Investigational Site, Torrance, California
  - Lyra Investigational Site, Boca Raton, Florida
  - Lyra Investigational Site, Boynton Beach, Florida
  - Lyra Investigational Site, Plantation, Florida
  - Lyra Investigational Site, Port Saint Lucie, Florida
  - Lyra Investigational Site, Chicago, Illinois
  - Lyra Investigational Site, Louisville, Kentucky
  - Lyra Investigational Site, Baltimore, Maryland
  - Lyra Investigational Site, New Hyde Park, New York
  - Lyra Investigational Site, New York, New York
  - Lyra Investigational Site, Winston-Salem, North Carolina
  - Lyra Investigational Site, Charleston, South Carolina
  - Lyra Investigational Site, Spartanburg, South Carolina
  - Lyra Investigational Site, Nashville, Tennessee
  - Lyra Investigational Site, Fort Worth, Texas
  - Lyra Investigational Site, Houston, Texas
  - Lyra Investigational Site, Mansfield, Texas
  - Lyra Investigational Site, San Antonio, Texas
  - Lyra Investigational Site, South Ogden, Utah
  - Lyra Investigational Site, Norfolk, Virginia
- Austria (4):
  - Lyra Investigational Site, Graz
  - Lyra Investigational Site, Klagenfurt
  - Lyra Investigational Site, Linz
  - Lyra Investigational Site, Vienna
- Czechia (5):
  - Lyra Investigational Site, Brno
  - Lyra Investigational Site, Hradec Králové
  - Lyra Investigational Site, Motol
  - Lyra Investigational Site, Olomouc
  - Lyra Investigational Site, Prague
- Poland (9):
  - Lyra Investigational Site, Bydgoszcz
  - Lyra Investigational Site, Elblag
  - Lyra Investigational Site, Katowice
  - Lyra Investigational Site, Krakow
  - Lyra Investigational Site, Krosno
  - Lyra Investigational Site, Lublin
  - Lyra Investigational Site, Nadarzyn
  - Lyra Investigational Site, Warsaw
  - Lyra Investigational Site, Wroclaw
- Spain (7):
  - Lyra Investigational Site, Barcelona
  - Lyra Investigational Site, Bilbao
  - Lyra Investigational Site, Cadiz
  - Lyra Investigational Site, Granada
  - Lyra Investigational Site, Madrid
  - Lyra Investigational Site, Navarro
  - Lyra Investigational Site, Santander

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Week 24 Treatment Period: 2:1 (LYR-210 to Sham) Randomization;
  Safety Extension Period: Sham participants received LYR-210; LYR-210 participants received LYR-210 or Sham (1:1)
Groups:
- LYR-210 - LYR-210: Repeat administration of LYR-210 at Week 24.
  Participants randomized to LYR-210 during the Week 24 Treatment Period received LYR-210 in the Safety Extension.
  Background therapy: Saline rinse
- LYR-210 - Sham: Crossover from LYR-210 to sham procedure control at Week 24.
  Participants randomized to LYR-210 during the Week 24 Treatment Period received sham procedure contol in the Safety Extension.
  Background therapy: Saline rinse
- Sham - LYR-210: Crossover from sham procedure control to LYR-210 at Week 24.
  Participants randomized to sham procedure contril during the Week 24 Treatment Period received LYR-210 in the Safety Extension.
  Background therapy: Saline rinse
Period: Week 24 Treatment Period
Arm/Group | LYR-210 | Sham Procedure Control | LYR-210 - LYR-210 | LYR-210 - Sham | Sham - LYR-210
Started | 130 | 66 | 0 | 0 | 0
Entered Extension | 84 | 52 | 0 | 0 | 0
Did Not Enter Extension | 40 | 14 | 0 | 0 | 0
Completed (Completed Week 24 Treatment) | 103 | 63 | 0 | 0 | 0
Not Completed | 27 | 3 | 0 | 0 | 0
Not completed — Treatment administration failure/procedure not attempted | 6 | 0 | 0 | 0 | 0
Not completed — Bilateral dislodgement | 13 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Other, not specified | 3 | 0 | 0 | 0 | 0
Period: Safety Extension Period
Arm/Group | LYR-210 | Sham Procedure Control | LYR-210 - LYR-210 | LYR-210 - Sham | Sham - LYR-210
Started | 0 | 0 | 42 | 42 | 52
Completed | 0 | 0 | 34 | 39 | 42
Not Completed | 0 | 0 | 8 | 3 | 10
Not completed — Treatment administration failure | 0 | 0 | 0 | 1 | 4
Not completed — Bilateral dislodgement | 0 | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | LYR-210 | Sham Procedure Control | Total
Number analyzed (Participants) | 124 | 66 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 58 | 165
  >=65 years | 17 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (13.65) | 45 (14.42) | 48 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 31 | 84
  Male | 71 | 35 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 22
  Not Hispanic or Latino | 111 | 57 | 168
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 111 | 54 | 165
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 3 | 1 | 4
  United States | 80 | 42 | 122
  Czechia | 9 | 1 | 10
  Poland | 28 | 20 | 48
  Spain | 4 | 2 | 6
BMI [Mean (Standard Deviation); unit: kg/m²] | 27.9 (5.63) | 27.4 (4.96) | 27.7 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFBL) in the 7-day Average Composite Score of 3 Cardinal Symptoms (3CS) in Participants Without Nasal Polyps.
Description: The 3CS are nasal blockage/obstruction/congestion, anterior/posterior nasal discharge, and facial pain/pressure. The diary is completed daily by study participants throughout the study. Each symptom/each question is rated on a 4-point (0-3) scale where 0= none/absent symptoms, 1=mild symptoms, 2=moderate symptoms, and 3=severe symptoms. The composite score of 3CS is the sum of the three cardinal symptom scores.
  The 3CS total score ranges from 0-9, with higher scores indicating worse symptoms.
Time Frame: 24 Weeks
Population: ITT Analysis Set Without Nasal Polyps
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LYR-210 | Sham Procedure Control
Number analyzed (Participants) | 101 | 54
score on a scale | -2.13 (2.172) | -2.06 (2.136)

2. Secondary Outcome: CFBL in the 7-day Average Composite Score of 3CS in All Participants at Week 24.
Description: as for outcome 1
Time Frame: Week 24
Population: ITT Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LYR-210 | Sham Procedure Control
Number analyzed (Participants) | 124 | 66
score on a scale | -2.35 (2.278) | -1.83 (2.104)

3. Secondary Outcome: CFBL in the 22-item Sino-Nasal Outcome Test (SNOT-22) Total Score at Week 24
Description: The SNOT-22 questionnaire is a 22-item disease-specific quality of life instrument. Each symptom is scored on a 6-point scale where 0 = no problem and 5 = problem as bad as it can be. The total SNOT-22 score is the sum of the 22 items and can range from 0 to 110 with higher scores indicating worse symptoms.
Time Frame: Week 24
Population: ITT Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LYR-210 | Sham Procedure Control
Number analyzed (Participants) | 124 | 66
score on a scale | -19.7 (21.67) | -15.7 (18.55)

4. Secondary Outcome: CFBL in the 3-D Volumetric CT Score at Week 20
Description: The percent opacification of the bilateral anterior and posterior ethmoids will be assessed by 3-D volumetric CT analysis at baseline and Week 20.
  A negative change from Baseline indicates improvement from Baseline.
Time Frame: Week 20
Population: ITT Analysis Set
Measure: Mean (Standard Deviation); unit: Percent ethmoid opacification
Arm/Group | LYR-210 | Sham Procedure Control
Number analyzed (Participants) | 124 | 66
Percent ethmoid opacification | -2.705 (10.9320) | -0.279 (9.9706)

5. Secondary Outcome: Participants With Rescue Treatments for CRS Through Week 24
Description: This endpoint is descriptively summarized per the prespecified plan. This includes participants that used systemic corticosteroid for any reason as well as participants that were recommended/underwent sinonasal surgery.
Time Frame: Week 24
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LYR-210 | Sham Procedure Control
Number analyzed (Participants) | 124 | 66
Participants | 12 | 7

ADVERSE EVENTS:
Time Frame: AEs are reported from the time the informed consent form is signed until completion of all follow-up visits, up to Week 52. Week 24 Treatment TEAEs: AEs that start on or after the LYR-210/Sham placement procedure but no later than 31 days after discontinuation of the first study treatment (up to 24 weeks). Extension Period TEAEs: AEs that start on or after the second placement procedure (Week 24) but no later than 31 days after discontinuation of second study treatment (up to Week 52).
Description: 190 participants successfully received treatment during the Week 24 Treatment Period. 6 participants who had a treatment administration failure are not included.
  131 participants successfully received study treatment during the Extension Period. 5 participants who had a treatment administration failure are not included.
Groups:
- LYR-210 up to 24 Weeks: Single administration of LYR-210 drug matrix (7500 μg)
  LYR-210: LYR-210 drug matrix (mometasone furoate)
  Background Therapy: Daily Saline Irrigation
- Sham Procedure Control up to 24 Weeks: Single mock administration procedure
  Sham procedure control: Sham procedure control
  Background Therapy: Daily Saline Irrigation
- LYR-210-LYR-210 Extension: Repeat administration of LYR-210 at Week 24
- LYR-210-Sham Extension: Crossover from LYR-210 to sham procedure control at Week 24
- Sham-LYR-210 Extension: Crossover from sham procedure control to LYR-210 at Week 24
Arm/Group | LYR-210 up to 24 Weeks | Sham Procedure Control up to 24 Weeks | LYR-210-LYR-210 Extension | LYR-210-Sham Extension | Sham-LYR-210 Extension
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/66 | 0/42 | 0/41 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/124 | 4/66 | 2/42 | 3/41 | 3/48
Other Adverse Events (participants affected / at risk) | 78/124 | 26/66 | 21/42 | 9/41 | 19/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYR-210 up to 24 Weeks (N=124) | Sham Procedure Control up to 24 Weeks (N=66) | LYR-210-LYR-210 Extension (N=42) | LYR-210-Sham Extension (N=41) | Sham-LYR-210 Extension (N=48)
Colonic Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical Device Site Joint Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYR-210 up to 24 Weeks (N=124) | Sham Procedure Control up to 24 Weeks (N=66) | LYR-210-LYR-210 Extension (N=42) | LYR-210-Sham Extension (N=41) | Sham-LYR-210 Extension (N=48)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 7 (8) | 6 (8) | 2 (2) | 4 (6)
Nasal Odour (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 0 (0) | 6 (7) | 0 (0) | 8 (10)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (11) | 10 (13) | 1 (1) | 1 (1) | 1 (1)
Chronis Sinusitis (Infections and infestations) | 14 (19) | 3 (4) | 6 (7) | 4 (5) | 4 (5)
COVID-19 (Infections and infestations) | 10 (10) | 4 (4) | 3 (3) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (11) | 6 (6) | 4 (4) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 13 (14) | 3 (4) | 4 (4) | 2 (3) | 3 (3)
Acute Sinusitis (Infections and infestations) | 14 (15) | 0 (0) | 2 (2) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except as approved by Sponsor, single center data will not be published before multicenter data, unless >1 year has elapsed since completion of the Study. PI may publish single center data provided that PI shall: i) provide a copy of the publication to Sponsor at least 60 days in advance of submission for publication; ii) delete Sponsor Confidential Information and make other reasonable changes; and iii) delay submission by up to 90 additional days to permit intellectual property filings.

DOCUMENTS (2):
  • Study Protocol (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT05219968/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT05219968/SAP_001.pdf